CLINICAL TRIAL: NCT00636805
Title: A Phase II Single Arm Trial of Palonosetron (PALO) for the Prevention of Acute and Delayed Chemotherapy Induced Nausea and Vomiting (CINV) in Malignant Glioma (MG) Patients Receiving Irinotecan in Combination With Bevacizumab
Brief Title: Aloxi for Prevention of Chemotherapy Induced Nausea and Vomiting in Malignant Glioma Patients Receiving Irinotecan With Bevacizumab
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was halted early after 63 subjects were enrolled due to slow accrual.
Sponsor: Duke University (Other)
Collaborators: Eisai Inc. (Industry); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00002273; P50NS020023 (NIH)
Record Dates: First submitted 2008-02-27; First posted 2008-03-14 (Estimated); Results first posted 2014-04-01 (Estimated); Last update posted 2014-04-01 (Estimated); Status verified 2014-03

CONDITIONS: Brain Cancer
Keywords: Aloxi; Brain Neoplasm, Primary; Brain Neoplasms, Malignant
MeSH Terms: conditions — Brain Neoplasms | interventions — Palonosetron; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Patient receives IV Aloxi
  Interventions: Drug: Palonosetron (Aloxi) and Dexamethasone

INTERVENTIONS:
Drug: Palonosetron (Aloxi) and Dexamethasone — single i.v. , dose of palonosetron 0.25 mg, and 10mg dexamethasone infused over 15 min, administered 30 min before the first dose Irinotecan and Bevacizumab chemotherapy.
  Other Names: Aloxi

SUMMARY:
1. Primary Objective:

   * To determine the efficacy and tolerability of palonosetron and dexamethasone in preventing acute CINV in brain tumor patients during the first 24 hours of receiving Irinotecan /Bevacizumab regimens.
2. Secondary Objective

   * To determine the safety and tolerability of palonosetron in brain tumor patients.
   * To determine the effects of glucocorticoid and anticonvulsants on the efficacy of palonosetron.
   * To determine the efficacy of palonosetron and dexamethasone in preventing delayed CINV in brain tumor patients during days 2-5.
   * To determine if patients receiving palonosetron have less fatigue than baseline.

DETAILED DESCRIPTION:
Before the patients receive the palonosetron, a physical exam and blood tests are performed to determine eligibility. If eligible and willing, subjects are given Palonosetron intravenously. Subjects are given the Palonosetron and Dexamethasone 30 minutes before the first dose of Irinotecan and Bevacizumab chemotherapy. The total expected duration of participation is 57 days. Subjects are also asked to complete 4 questionnaires about nausea and vomiting, as well as daily functioning and fatigue. Subjects are asked to complete these questionnaires before starting chemotherapy, the day of starting chemotherapy and for the next 4 days after receiving chemotherapy, for a total of 6 times. Subjects are asked to complete this set of questionnaires each of the 3 times that they receive chemotherapy during the 6-week treatment cycle.

The other treatments subjects would normally receive for their brain tumor and their routine care are not affected by the study.

ELIGIBILITY:
Inclusion Criteria:

In order to be included in the study, patients must meet all of the following criteria:

* Patients must have histologically confirmed diagnosis of primary malignant glioma (glioblastoma multiforme, gliosarcoma or anaplastic astrocytoma, or anaplastic oligodendroglioma) who are either chemotherapy naïve or non-naïve and scheduled to receive Irinotecan/Bevacizumab chemotherapy.
* Patients with recurrent disease whose diagnostic pathology confirmed malignant glioma (glioblastoma multiforme, gliosarcoma or anaplastic astrocytoma, or anaplastic oligodendroglioma) will not need re-biopsy.
* Age > or = 18 years.
* Patient is scheduled to receive Irinotecan/Bevacizumab chemotherapy every 2 weeks for one complete 6-week cycle.
* An interval of at least 6 weeks between prior surgical resection and study enrollment.
* An interval of at least 4 weeks between prior radiotherapy and enrollment on this protocol unless there is unequivocal evidence of tumor progression after radiotherapy or chemotherapy.
* The lab values following the prior chemotherapy must return within normal limits prior to study enrollment.
* Karnofsky > 60%.
* Hematocrit > 29%, absolute neutrophil count (ANC) > 1,500 cells/*l, platelets > 125,000 cells/*l.
* Serum creatinine < 1.5 mg/dl, serum glutamic-oxaloacetic transaminase (SGOT) and bilirubin < 1.5 times upper limit of normal.
* Patients on corticosteroids must be on a stable dose for 1 week prior to entry, and the dose should not be escalated over entry dose level, if clinically possible.
* Signed consent form approved by the Institutional Review Board prior to patient entry.
* No evidence of hemorrhage on the baseline MRI or CT scan.
* If sexually active, patients will take contraceptive measures for the duration of the treatments.

Exclusion Criteria:

Patients are excluded from this study if they meet any of the following criteria:

* Inability or unwillingness to understand or cooperate with study procedures.
* Received any intravenous drug with potential anti-emetic effect within 24 hours prior to the start of study-designated chemotherapeutic agent or be scheduled to receive any drug of this type (with the exception of administration of the palonosetron/dexamethasone infusion solution) at any time during the trial, including the following:
* 5 HT3 receptor antagonists;
* Dopamine receptor antagonists (metoclopramide);
* Phenothiazine anti-emetics (prochlorperazine, thiethylperazine and perphenazine);
* Diphenhydramine, scopolamine, chlorpheniramine maleate, trimethobenzamide. Diphenhydramine will be allowed if given for prophylactic treatment of hypersensitivity reactions associated with the administration of taxanes;
* Haloperidol, droperidol, tetrahydrocannabinol, or nabilone; and
* Any systemic corticosteroid (hydrocortisone, methylprednisolone, prednisone). Topical or inhaled preparations are allowed;
* Previous participation in any clinical trial involving palonosetron (RS-25259 of Syntex).
* Any vomiting, retching or NCI Common Toxicity Criteria version 3.0 grade 2-4 nausea (see Appendix 8.6) in the 24 hours preceding chemotherapy.
* Ongoing vomiting from any organic etiology.
* Will receive radiotherapy of upper abdomen or cranium within one week prior to or during the study.
* Received palonosetron within 14 days prior to study enrollment (AloxiTM).
* Evidence of central nervous system (CNS) hemorrhage on baseline MRI on CT scan.
* Co -medication that may interfere with study results; e.g. immuno-suppressive agents other than corticosteroids.
* Prophylactic medication for the prevention of nausea and vomiting 24 hours prior to the start of chemotherapy through 120 hours after the initiation of chemotherapy on Study Day 1 (Study Day 6) is prohibited, with the exception of the study drug. Corticosteroids will be allowed for treatment of cerebral swelling. Diphenhydramine will be allowed only if given for prophylactic treatment of hypersensitivity reactions associated with the administration of taxanes, as per the package insert for these agents. Rescue medication for treatment of nausea and vomiting is permitted after chemotherapy at the discretion of the investigator. The agent, dose, and time of administration will be recorded in the patient diary.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2008-05; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Lou Affronti, RN, MSN, ANP, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Patient Receives IV Aloxi: Patient receives IV Aloxi
  Palonosetron (Aloxi) and Dexamethasone: single i.v. , dose of palonosetron 0.25 mg, and 10mg dexamethasone infused over 15 min, administered 30 min before the first dose Irinotecan and Bevacizumab chemotherapy.
Period: Overall Study
Arm/Group | Patient Receives IV Aloxi
Started | 63
Completed | 63
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patient Receives IV Aloxi
Number analyzed (Participants) | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.2 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 42

OUTCOME MEASURES:

1. Primary Outcome: Acute CINV (Chemotherapy Induced Nausea and Vomiting) CR (Complete Response) Rate
Description: Acute Chemotherapy-Induced Nausea and Vomiting (CINV) complete response (CR) rate is defined as the percentage of patients who do not have an emetic episode or use antiemetic rescue medication during the first 24 hours following chemotherapy of the first cycle of treatment.
Time Frame: first 24 hours of the first week of chemotherapy
Population: Intent-to-treat; 11 patients did not complete the study measure for day 1 of the first week of chemotherapy
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Patient Receives IV Aloxi
Number analyzed (Participants) | 52
percentage of participants | 62 [47 to 75]

2. Secondary Outcome: Acute Chemotherapy-Induced Nausea and Vomiting (CINV) Complete Response (CR) Rate by Corticosteroid Use at Baseline
Description: as for outcome 1
Time Frame: Day 1 of the first week of chemotherapy
Population: Intent-to-treat; 11 patients did not complete the study measure for day 1 of the first week of chemotherapy
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Patient Receives IV Aloxi
Number analyzed (Participants) | 52
percentage of participants
  corticosteroid used at baseline | 68 [43 to 87]
  no corticosteroid used at baseline | 58 [39 to 75]

3. Secondary Outcome: Acute Chemotherapy-Induced Nausea and Vomiting (CINV) Complete Response (CR) Rate by Anticoagulant Use at Baseline
Description: as for outcome 1
Time Frame: Day 1 of the first week of chemotherapy
Population: Intent-to-treat; 11 patients did not complete the study measure for day 1 of the first week of chemotherapy
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Patient Receives IV Aloxi
Number analyzed (Participants) | 52
percentage of participants
  anticoagulant used at baseline | 61 [43 to 77]
  no anticoagulant used at baseline | 63 [35 to 85]

4. Secondary Outcome: Delayed Chemotherapy-Induced Nausea and Vomiting (CINV) Complete Response (CR) Rate
Description: Delayed Chemotherapy-Induced Nausea and Vomiting (CINV) complete response (CR) rate is defined as the percentage of patients who do not have an emetic episode or use antiemetic rescue medication during days 2 through 5 of chemotherapy treatment during the first cycle of treatment
Time Frame: Days 2-5 of the first week of chemotherapy
Population: Intent-to-treat; 10 patients did not complete the study measure for days 2-5 of the first week of chemotherapy
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Patient Receives IV Aloxi
Number analyzed (Participants) | 53
percentage of participants | 62 [48 to 75]

5. Secondary Outcome: Percentage of Patients With ≥ Grade 3, Treatment-related Toxicities
Description: Percentage of patients with ≥ grade 3, treatment-related toxicities using the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0.
Time Frame: 6 weeks
Measure: Number; unit: participants
Arm/Group | Patient Receives IV Aloxi
Number analyzed (Participants) | 63
participants | 0

6. Secondary Outcome: Overall Mean Change in the Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Score From Baseline to Day 5 of the First Week of Chemotherapy
Description: Overall mean change in the Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue score from baseline to day 5 of the first week of chemotherapy. The FACIT-Fatigue is a 13-item validated questionnaire assessing the impact of fatigue on an individual's quality of life. The raw score range is 0-52 with higher scores indicating better quality of life. The mean change from baseline to day 5 was calculated by subtracting the baseline score from mean of the day 1-5 scores, thus a negative mean change represents worsening in quality of life due to fatigue.
Time Frame: Baseline through day 5 of the first week of chemotherapy
Population: Intent-to-treat; 16 patients did not complete the study measure at baseline or on day 5 of the first week of chemotherapy
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Patient Receives IV Aloxi
Number analyzed (Participants) | 47
units on a scale | -3.5 [-6.1 to -0.9]

7. Secondary Outcome: Overall Mean Change in the Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Score From Baseline to Day 5 of the First Week of Chemotherapy by Acute Chemotherapy-Induced Nausea and Vomiting (CINV) Complete Response (CR)
Description: Overall mean change in the Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue score from baseline to day 5 of the first week of chemotherapy. The FACIT-Fatigue is a 13-item validated questionnaire assessing the impact of fatigue on an individual's quality of life. The raw score range is 0-52 with higher scores indicating better quality of life. The mean change from baseline to day 5 was calculated by subtracting the baseline score from the mean of the day 1-5 scores, thus a negative mean change represents worsening in quality of life due to fatigue. Acute CINV complete response (CR) is defined as not having an emetic episode or any use of antiemetic rescue medication during the first 24 hours following chemotherapy of the first cycle of treatment.
Time Frame: Baseline through day 5 of the first week of chemotherapy
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Patient Receives IV Aloxi
Number analyzed (Participants) | 47
units on a scale
  CR | -3.5 [-6.4 to -0.6]
  Not CR | -3.3 [-8.8 to 2.2]

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: The adverse events for this study were collected using Common Terminology Criteria for Adverse Events (CTCAE) version 3.0.
Arm/Group | Patient Receives IV Aloxi
Serious Adverse Events (participants affected / at risk) | 3/63
Other Adverse Events (participants affected / at risk) | 51/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patient Receives IV Aloxi (N=63)
White blood cell decreased (Investigations) | 1
Fatigue (General disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Infection - Other (Specify, CSF) (Infections and infestations) | 1
Infections and infestations (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Thromboembolic event (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patient Receives IV Aloxi (N=63)
Anemia (Blood and lymphatic system disorders) | 1
White blood cell decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 3
Fatigue (General disorders) | 20
Insomnia (Psychiatric disorders) | 18
Weight loss (Investigations) | 7
Burn (Injury, poisoning and procedural complications) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4
Rash acneiform (Skin and subcutaneous tissue disorders) | 3
Anorexia (Metabolism and nutrition disorders) | 11
Constipation (Gastrointestinal disorders) | 16
Diarrhea (Gastrointestinal disorders) | 20
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 2
Mucositis (Gastrointestinal disorders) | 10
Mucositis oral (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 24
Esophageal ulcer (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 10
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Infections and infestations - Other, specify (Infections and infestations) | 7
Bladder infection (Infections and infestations) | 1
pneumonia (Infections and infestations) | 1
Proteinuria (Renal and urinary disorders) | 1
Ataxia (Nervous system disorders) | 15
Cognitive disturbance (Nervous system disorders) | 19
Confusion (Nervous system disorders) | 18
Dizziness (Nervous system disorders) | 13
Memory impairment (Nervous system disorders) | 16
Mood alteration (Nervous system disorders) | 16
Peripheral motor neuropathy (Nervous system disorders) | 19
Peripheral sensory neuropathy (Nervous system disorders) | 6
Seizure (Nervous system disorders) | 10
Depressed level of consciousness (Nervous system disorders) | 23
Dysphasia (Nervous system disorders) | 9
Tremor (Nervous system disorders) | 11
Blurred vision (Eye disorders) | 12
Headache (Nervous system disorders) | 13
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8
Urinary incontinence (Renal and urinary disorders) | 2
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research site shall provide MGI copies of publication at least 30 days prior to submission to allow MGI to protect its copyrights, to determine any Confidential Information (CI) and to check for technical correctness. Site shall consider any MGI comments and delete any CI requested by MGI, unless CI removal changes accuracy or interpretation of results, in which case site and MGI will discuss timing of submission. MGI may request delay of up to 60 days to protect its copyright or patent rights.